CLINICAL TRIAL: NCT00286013
Title: Feasibility of Radiotherapy and Concomitant Gemcitabine and Oxaliplatin in Locally Advanced Pancreatic Cancer and Distal Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/196
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Locally Advanced and Unresectable, But Non-metastatic Pancreatic Adenocarcinoma or Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Association of gemcitabine, oxaliplatin and radiotherapy

SUMMARY:
The aim of the study is to evaluate the feasibility defined as overall tolerance and toxicity as well as relative dose-intensity and cumulative dose delivered, of an association ofgemcitabine, oxaliplatin and radiotherapy in patients with locally advanced and unresectable, but non-metastatic pancreatic adenocarcinoma or cholangiocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven and unresectable adenocarcinoma of the pancreas or cholangiocarcinoma with no evidence of metastatic disease
* WHO performance status of 0 or 1
* Complete recovrey from surgery in case an enteric and/or biliary tract by-pass operation has been performed
* Maximum delay after surgery: 8 weeks
* No previous or co-existent malignant disease except non melanoma skin cancers and adequately treated cervic carcinoma in situ
* Adequate bon marrow reserve
* No previous chemotherapy or radiotherapy
* Expected survival > 6 months

Exclusion Criteria:

* Active infection
* Metastatic disease
* Inadequate liver function after derivative surgery
* Inadequate renal function
* Pregnancy, breast feeding
* Use of any other investigational agent in the month before enrollment
* Patients with grade 2 or more neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-05-01 (Actual); Primary Completion 2006-05-31 (Actual); Study Completion 2008-07-22 (Actual)

PRIMARY OUTCOMES:
Feasibility
Tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Marc Peeters, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (4):
- Belgium (4):
  - Erasme University Hospital, Brussels
  - Jules Bordet Institute, Brussels
  - University Hospital Ghent, Ghent
  - CHU Sart-Tilman, Liège

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be